CLINICAL TRIAL: NCT03319667
Title: A Phase 3 Randomized, Open-label, Multicenter Study Assessing the Clinical Benefit of Isatuximab (SAR650984) in Combination With Bortezomib (Velcade®), Lenalidomide and Dexamethasone Versus Bortezomib, Lenalidomide and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Not Eligible for Transplant
Brief Title: A Study to Investigate the Clinical Benefit of Isatuximab in Combination With Bortezomib, Lenalidomide and Dexamethasone in Adults With Newly Diagnosed Multiple Myeloma Not Eligible for Transplant
Acronym: IMROZ
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFC12522; U1111-1194-2121 (Registry Identifier: ICTRP); 2024-514417-34 (Registry Identifier: CTIS); 2017-002238-21 (EudraCT Number)
Record Dates: First submitted 2017-09-18; First posted 2017-10-24 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Parallel and crossover
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Isatuximab/Bortezomib/Lenalidomide/Dexamethasone = IVRd arm (Experimental): 1. Induction treatment with 4x6-week cycles with intravenous (IV) isatuximab + subcutaneous (SC) bortezomib + oral lenalidomide + IV or oral dexamethasone
  2. Continuous treatment with 4-week cycles with IV isatuximab + oral lenalidomide + IV or oral dexamethasone
  Interventions: Drug: Isatuximab SAR650984; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Bortezomib/Lenalidomide/Dexamethasone = VRd arm (Active Comparator): 1. Induction treatment with 4x6-week cycles with SC bortezomib + oral lenalidomide + IV or oral dexamethasone
  2. Continuous treatment with 4-week cycles with oral lenalidomide + IV or oral dexamethasone
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Isatuximab/Lenalidomide/Dexamethasone = IRd crossover arm (Other): 4-weeks cycles with IV isatuximab + oral lenalidomide + IV or oral dexamethasone
  Interventions: Drug: Isatuximab SAR650984; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form: Solution for infusion
  Route of administration: Intravenous (IV)
  Other Names: Sarclisa
  Arms: Isatuximab/Bortezomib/Lenalidomide/Dexamethasone = IVRd arm; Isatuximab/Lenalidomide/Dexamethasone = IRd crossover arm
Drug: Bortezomib — Pharmaceutical form: Lyophilized powder for injection
  Route of administration: Subcutaneous
  Other Names: Velcade®
  Arms: Bortezomib/Lenalidomide/Dexamethasone = VRd arm; Isatuximab/Bortezomib/Lenalidomide/Dexamethasone = IVRd arm
Drug: Lenalidomide — Pharmaceutical form: Capsules
  Route of administration: Oral
Drug: Dexamethasone — Pharmaceutical form: Tablets, ampoules or vials for injection
  Route of administration: Oral/Intravenous

SUMMARY:
Primary Objective:

-To demonstrate the benefit of isatuximab in combination with bortezomib, lenalidomide, and dexamethasone in the prolongation of progression free survival (PFS) as compared to bortezomib, lenalidomide, and dexamethasone, in participants with newly diagnosed multiple myeloma (NDMM) not eligible for transplant.

Secondary Objectives:

* To evaluate in both randomized (isatuximab, bortezomib, lenalidomide and dexamethasone combination (IVRd) and bortezomib, lenalidomide and dexamethasone combination (VRd)) arms:
* Complete response (CR) rate, as defined by the International Myeloma Working Group (IMWG) criteria.
* Minimal residual disease (MRD) negativity rate in participants with CR.
* Very good partial response or better rate, as defined by the IMWG criteria.
* Overall survival (OS).
* To evaluate the overall response rate (ORR) as per IMWG criteria.
* To evaluate the time to progression (TTP) overall and by MRD status.
* To evaluate PFS by MRD status.
* To evaluate the duration of response (DOR) overall and by MRD status.
* To evaluate time to first response (TT1R).
* To evaluate time to best response (TTBR).
* To evaluate progression-free survival on next line of therapy (PFS2).
* To evaluate the sustained MRD negativity >12 months rate.
* To evaluate safety.
* To determine the pharmacokinetic (PK) profile of isatuximab in combination with bortezomib, lenalidomide, and dexamethasone (IVRd arm only).
* To evaluate the immunogenicity of isatuximab in participants receiving isatuximab (IVRd and crossover arms).
* To assess disease-specific and generic health-related quality of life (HRQL), disease and treatment-related symptoms, health state utility, and health status.

DETAILED DESCRIPTION:
The duration of the study for each participant will include a screening period of up to 4 weeks, an induction period of 24 weeks (4 cycles with a duration of 42 ± 3 days), a continuous treatment period and a crossover period (when applicable). The cycle duration is 28 ± 3 days during the continuous treatment and crossover periods.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria :

* Multiple myeloma (IMWG criteria).
* Newly diagnosed multiple myeloma not eligible for transplant due to age (≥ 65 years) or participants < 65 years with comorbidities impacting possibility of transplant.
* Evidence of measurable disease.
* Written informed consent.

Exclusion criteria:

* Age < 18 years.
* Prior treatment for multiple myeloma.
* Any other prior or ongoing disease/health conditions incompatible with the study objectives.
* Organ function values not met.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ( PS) > 2.
* Hypersensitivity to the study medications.
* Pregnant, breastfeeding, or woman of child bearing potential unwilling to use recommended contraception methods.
* Male participants who disagree to follow the study contraceptive counseling.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 100 months after the First Participant In (FPI)
  Defined as the time from the date of randomization to the date of first documentation of progression disease (PD) as determined by the independent review committee (IRC) or the date of death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Complete response rate (CR) | Up to approximately 100 months after the FPI
  Defined as the proportion of participants with CR and stringent complete response (sCR) as assessed by the IRC using the IMWG criteria.
Minimal residual disease (MRD) negativity rate for participants with CR | Up to approximately 100 months after the FPI
  Proportion of participants with CR for whom MRD measurement is negative
Very good partial response (VGPR) or better rate | Up to approximately 100 months after the FPI
  Proportion of participants with sCR, CR and VGPR as assessed by the IRC using the International Myeloma Working Group (IMWG) criteria
Overall survival (OS) | Up to approximately 110 months after the FPI
  Defined as the time from the date of randomization to death from any cause
Overall response rate (ORR) | Up to approximately 100 months after the FPI assessment
  Proportion of participants with best overall response (BOR) recorded as sCR, CR, VGPR, or partial response (PR) as assessed by the IRC using the IMWG criteria
Time to progression (TTP) | Up to approximately 100 months after FPI
  Defined as the time from randomization to date of first documentation of PD as assessed by the IRC using the IMWG criteria
Duration of response (DOR) | Up to approximately 100 months after the FPI
  Defined as the time from date of first IRC determined response to date of first IRC PD or death, whichever occurs first for participants achieving sCR, CR, VGPR, or PR
Time to first response (TT1R) | Up to approximately 100 months after the FPI
  Time from randomization to the first IRC determined response (PR or better) that is subsequently confirmed
Time to best response (TTBR) | Up to approximately 100 months after the FPI
  Defined as the time from randomization to the date of first occurrence of IRC determined best response (PR or better) that is subsequently confirmed
PFS on next line of therapy (PFS2) | Up to approximately 110 months after the FPI
  Defined as the time from randomization to the date of first documentation of disease progression (as assessed by investigator) after initiation of further anti-myeloma treatment, or death from any cause, whichever occurs first
PFS in MRD negative participants | Up to approximately 100 months after the FPI
  Defined as the time from the date of randomization to the date of first documentation of PD or the date of death from any cause, whichever comes first in MRD negative participants
Sustained MRD negativity ≥12 months rate | Up to approximately 100 months after the FPI
  Defined as the proportion of participants with the maintenance of MRD negativity confirmed ≥12 months apart with no MRD positive test in between.
Adverse Events | Up to 30 days after end of treatment (EOT) visit
  Treatment-emergent adverse events/serious adverse events (TEAEs/SAEs) including infusion associated reactions (IARs), second primary malignancies, laboratory parameters, vital signs, weight, ECOG PS, and findings from physical examination
Assessment of PK parameter: Ctrough | Cycle 1 Day 8/Day 15/Day 29 (pre-dose) and Day 1 (pre-dose) of Cycle 2, 3, 4, 5, 6, 7, 8, 9 and 10 (Duration of each cycle for Cycles 1-4: 6 weeks; Duration of each cycle for Cycles 5-10: 4 weeks)
  Isatuximab: Pre-dose plasma isatuximab concentration (Ctrough)
Immunogenicity | Up to approximately 100 months after the FPI
  Presence of anti-drug antibodies against isatuximab
participants reported outcome (PRO): QLQ-C30 | Up to approximately 100 months after the FPI
  Disease-specific HRQL will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) core quality of life questionnaire (QLQ-C30)
PRO: QLQ-MY20 | Up to approximately 100 months after the FPI
  Disease- and treatment-related quality of life will be assessed using the EORTC myeloma module (QLQ-MY20) questionnaire
PRO: EQ-5D-5L | Up to approximately 100 months after the FPI
  Health state utility and health status will be assessed using the European Quality of Life Group questionnaire with 5 dimensions and 5 levels per dimension (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (104):
- United States (5):
  - Investigational Site Number: 8400006, Fort Myers, Florida
  - Investigational Site Number: 8400004, St. Petersburg, Florida
  - Investigational Site Number: 8400007, Kansas City, Missouri
  - Investigational Site Number: 8400005, Nashville, Tennessee
  - Investigational Site Number: 8400001, Houston, Texas
- Australia (8):
  - Investigational Site Number : 0360003, Liverpool, New South Wales
  - Investigational Site Number : 0360001, Waratah, New South Wales
  - Investigational Site Number : 0360002, Wollongong, New South Wales
  - Investigational Site Number : 0360007, South Brisbane, Queensland
  - Investigational Site Number : 0360005, Clayton, Victoria
  - Investigational Site Number : 0360004, Heidelberg West, Victoria
  - Investigational Site Number : 0360006, Nedlands, Western Australia
  - Investigational Site Number : 0360008, West Perth, Western Australia
- Investigational Site Number : 0560001, Liège, Belgium
- China (13):
  - Investigational Site Number : 1560002, Beijing
  - Investigational Site Number : 1560003, Beijing
  - Investigational Site Number : 1560008, Changchun
  - Investigational Site Number : 1560007, Fuzhou
  - Investigational Site Number : 1560009, Guangzhou
  - Investigational Site Number : 1560006, Guangzhou
  - Investigational Site Number : 1560005, Hangzhou
  - Investigational Site Number : 1560014, Hangzhou
  - Investigational Site Number : 1560004, Nanjing
  - Investigational Site Number : 1560013, Shanghai
  - Investigational Site Number : 1560011, Shenyang
  - Investigational Site Number : 1560001, Tianjin
  - Investigational Site Number : 1560012, Wuhan
- Czechia (6):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030007, Hradec Králové
  - Investigational Site Number : 2030004, Olomouc
  - Investigational Site Number : 2030003, Ostrava - Poruba
  - Investigational Site Number : 2030006, Pilsen
  - Investigational Site Number : 2030001, Prague
- Denmark (3):
  - Investigational Site Number : 2080002, Aalborg
  - Investigational Site Number : 2080003, Aarhus N
  - Investigational Site Number : 2080004, Odense C
- France (12):
  - Investigational Site Number : 2500011, Bayonne
  - Investigational Site Number : 2500007, Caen
  - Investigational Site Number : 2500009, Dijon
  - Investigational Site Number : 2500008, La Roche-sur-Yon
  - Investigational Site Number : 2500001, Lille
  - Investigational Site Number : 2500003, Nantes
  - Investigational Site Number : 2500012, Paris
  - Investigational Site Number : 2500002, Pessac
  - Investigational Site Number : 2500006, Pierre-Bénite
  - Investigational Site Number : 2500005, Poitiers
  - Investigational Site Number : 2500004, Toulouse
  - Investigational Site Number : 2500010, Vandœuvre-lès-Nancy
- Germany (4):
  - Investigational Site Number : 2760003, Berlin
  - Investigational Site Number : 2760004, Frankfurt am Main
  - Investigational Site Number : 2760001, Heidelberg
  - Investigational Site Number : 2760005, Tübingen
- Greece (3):
  - Investigational Site Number : 3000003, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Thessaloniki
- Italy (5):
  - Investigational Site Number : 3800005, Ancona
  - Investigational Site Number : 3800003, Bergamo
  - Investigational Site Number : 3800001, Bologna
  - Investigational Site Number : 3800004, Brescia
  - Investigational Site Number : 3800002, Torino
- Japan (10):
  - Investigational Site Number : 3920007, Nagoya, Aichi-ken
  - Investigational Site Number : 3920004, Higashiibaraki-gun, Ibaraki
  - Investigational Site Number : 3920008, Konan-ku, Yokohama-shi, Kanagawa
  - Investigational Site Number : 3920003, Kumamoto, Kumamoto
  - Investigational Site Number : 3920009, Sendai, Miyagi
  - Investigational Site Number : 3920005, Okayama, Okayama-ken
  - Investigational Site Number : 3920006, Sunto-gun, Shizuoka
  - Investigational Site Number : 3920001, Shibuya-ku, Tokyo
  - Investigational Site Number : 3920002, Shinjuku-ku, Tokyo
  - Investigational Site Number : 3920010, Yamagata
- Lithuania (2):
  - Investigational Site Number : 4400002, Klaipėda
  - Investigational Site Number : 4400001, Vilnius
- Investigational Site Number : 4840001, Monterrey, Nuevo León, Mexico
- New Zealand (3):
  - Investigational Site Number : 5540002, Takapuna, Auckland
  - Investigational Site Number : 5540003, Hamilton, Waikato Region
  - Investigational Site Number : 5540001, Auckland
- Poland (4):
  - Investigational Site Number : 6160004, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160003, Lodz, Lódzkie
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160002, Gdansk, Pomeranian Voivodeship
- Portugal (5):
  - Investigational Site Number : 6200002, Braga
  - Investigational Site Number : 6200006, Coimbra
  - Investigational Site Number : 6200001, Lisbon
  - Investigational Site Number : 6200005, Porto
  - Investigational Site Number : 6200003, Porto
- Russia (2):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430002, Moscow
- Spain (4):
  - Investigational Site Number : 7240005, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240001, Murcia
- Sweden (2):
  - Investigational Site Number : 7520002, Lund
  - Investigational Site Number : 7520001, Stockholm
- Taiwan (3):
  - Investigational Site Number : 1580003, Changhua
  - Investigational Site Number : 1580002, Taichung
  - Investigational Site Number : 1580001, Taipei
- Turkey (Türkiye) (8):
  - Investigational Site Number : 7920006, Adana
  - Investigational Site Number : 7920007, Ankara
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920004, Izmir
  - Investigational Site Number : 7920003, Izmir
  - Investigational Site Number : 7920005, Kayseri
  - Investigational Site Number : 7920008, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Manier S, Dimopoulos MA, Leleu XP, Moreau P, Cavo M, Goldschmidt H, Orlowski RZ, Tron M, Tekle C, Bregeault MF, Shafer AT, Beksac M, Facon T. Isatuximab plus bortezomib, lenalidomide, and dexamethasone for transplant-ineligible newly diagnosed multiple myeloma patients: a frailty subgroup analysis of the IMROZ trial. Haematologica. 2025 Sep 1;110(9):2139-2150. doi: 10.3324/haematol.2024.287200. Epub 2025 Mar 20. PMID 40109195
- [Derived] Facon T, Dimopoulos MA, Leleu XP, Beksac M, Pour L, Hajek R, Liu Z, Minarik J, Moreau P, Romejko-Jarosinska J, Spicka I, Vorobyev VI, Besemer B, Ishida T, Janowski W, Kalayoglu-Besisik S, Parmar G, Robak P, Zamagni E, Goldschmidt H, Martin TG, Manier S, Mohty M, Oprea C, Bregeault MF, Mace S, Berthou C, Bregman D, Klippel Z, Orlowski RZ; IMROZ Study Group. Isatuximab, Bortezomib, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2024 Oct 31;391(17):1597-1609. doi: 10.1056/NEJMoa2400712. Epub 2024 Jun 3. PMID 38832972
- [Derived] Thoren K, Menad S, Nouadje G, Mace S. Isatuximab-Specific Immunofixation Electrophoresis Assay to Remove Interference in Serum M-Protein Measurement in Patients with Multiple Myeloma. J Appl Lab Med. 2024 Jul 1;9(4):661-671. doi: 10.1093/jalm/jfae028. PMID 38573925